CLINICAL TRIAL: NCT05806515
Title: S2210 A Phase II Study of Neoadjuvant Carboplatin for Localized, High Risk Prostate Cancer With Germline BRCA1/2 Mutations
Brief Title: Carboplatin Chemotherapy Before Surgery for People With High-Risk Prostate Cancer and an Inherited BRCA1 or BRCA2 Gene Mutation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2210; NCI-2023-02356 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2210 (Other: SWOG); S2210 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma; Stage IIIB Prostate Cancer AJCC v8; Stage IIIC Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Specimen Handling; Carboplatin; X-Rays; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (carboplatin) (Experimental): Patients receive carboplatin IV on study. Patients then undergo surgery on study. Patients who experience PSA progression after surgery undergo CT or MRI of the abdomen and pelvis, CT of the chest or chest X-ray, or PSMA-PET throughout the trial. Patients also undergo collection of blood samples throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Chest Radiography; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: PSMA PET Scan; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Chest Radiography — Undergo chest X-ray
  Other Names: Chest X-ray
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: PSMA PET Scan — Undergo PSMA PET
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Procedure: Surgical Procedure — Undergo surgery
  Other Names: Operation; Surgery; Surgery Type; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase II trial tests how well carboplatin before surgery works in treating patients with high-risk prostate cancer and an inherited BRCA1 or BRCA2 gene mutation. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping, or slowing the growth of tumor cells. Giving carboplatin before surgery may shrink tumors in patients with high-risk prostate cancer with BRCA1 and BRCA2 gene mutations.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the pathologic complete response rate at prostatectomy in patients with localized high-risk prostate cancer with germline BRCA2 or BRCA1 mutations who are treated with neoadjuvant carboplatin by central review of source documents.

SECONDARY OBJECTIVES:

I. To evaluate prostate specific antigen (PSA) progression-free survival post-prostatectomy over the duration of follow-up and specifically, at the 3-year landmark.

II. To evaluate metastases free survival and overall survival. III. To evaluate the frequency and severity of toxicities of neoadjuvant carboplatin followed by radical prostatectomy.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

Patients receive carboplatin intravenously (IV) on study. Patients then undergo surgery on study. Patients who experience PSA progression after surgery undergo computed tomography (CT) or magnetic resonance imaging (MRI) of the abdomen and pelvis, CT of the chest or chest X-ray, or prostate-specific membrane antigen (PSMA)-positron emission tomography (PET) throughout the trial. Patients also undergo collection of blood samples throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologic diagnosis of prostate adenocarcinoma
* Participant must have high or very high-risk disease defined by at least one of the following:

  * cT3a - cT4x
  * Grade group 4 or 5 (Gleason sum 8-10)
  * PSA > 20 ng/mL prior to registration
* Participant must have documented evidence of germline mutation (pathogenic/likely pathogenic variant) in BRCA2 or BRCA1 through testing in a Clinical Laboratory Improvement Act (CLIA)-certified lab

  * NOTE: Local lab report is sufficient for eligibility
* Participant may have initiated gonadotrophin releasing hormone (gnRH) agonist, gnRH antagonist, oral anti-androgen (e.g. bicalutamide, nilutamide, flutamide), or other agent intended to treat prostate cancer prior to registration. The effectiveness of the current depot of such treatment must not extend beyond 1 month after study registration. Agents listed above cannot be started after participant registration
* Participant must be >= 18 years old
* Participant must have Zubrod performance status of 0-2
* Participant must have a complete medical history and physical exam within 28 days prior to registration
* Absolute neutrophil count >= 1.5 x 10^3/uL (within 28 days prior to registration)
* Platelets >= 100 x 10^3/uL (within 28 days prior to registration)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x institutional upper limit of normal (ULN) (within 28 days prior to registration)
* Participant must have a serum creatinine =< the institutional upper limit of normal (IULN) OR measured OR calculated creatinine clearance >= 50 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 28 days prior to registration
* Participant must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification within 28 days prior to registration. To be eligible for this trial, participants must be class 2B or better
* Participant with known human immunodeficiency virus (HIV)-infection must be receiving anti-retroviral therapy and have an undetectable viral load test within 6 months prior to registration
* Participant with history of chronic hepatitis B virus (HBV) infection must have undetectable HBV viral load on suppressive therapy within in 28 days prior to registration
* Participant with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment must have an undetectable HCV viral load within in 28 days prior to registration
* Participants who are of reproductive potential must have agreed to use an effective contraceptive method with details provided as a part of the consent process. A person who has semen likely to contain sperm is considered to be of "reproductive potential." In addition to routine contraceptive methods, "effective contraception" also includes refraining from sexual activity that might result in pregnancy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) including vasectomy with testing showing no sperm in the semen
* Prior to registration, participant must have had a urologic consult and be deemed a surgical candidate with known sites of disease deemed by the urologist to be potentially resectable
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* NOTE: As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines
  * For participants with impaired decision-making capabilities, legally authorized representatives may sign and give informed consent on behalf of study participants in accordance with applicable federal, local, and Central Institutional Review Board (CIRB) regulations
  * As part of the registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Exclusion Criteria:

* Participant must not have evidence of distant metastatic disease by conventional imaging within 90 days prior to registration

  * NOTE: cN1 detected only by PSMA-PET is permitted if urologist deems sites of disease to be potentially completely resectable
* Participant must not have received prior radiation therapy (RT) to the pelvic region
* Participant must not have a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) has the potential to interfere with the safety or efficacy assessment of protocol treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response after neoadjuvant carboplatin | Up to 5 years
  A two-stage design will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Heather H Cheng, Principal Investigator — SWOG Cancer Research Network
Locations (133):
- United States (133):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mercy Cancer Center �� Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Providence Queen of The Valley, Napa, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Providence Medical Foundation - Santa Rosa, Santa Rosa, California
  - Providence Santa Rosa Memorial Hospital, Santa Rosa, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Garnet Health Medical Center, Middletown, New York
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - FHCC South Lake Union, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming